



## MOTHER'S CONSENT FORM

Please initial Study no. ..... all boxes **GENERAL STATEMENTS** YES NO 1. I can confirm that I have read and understood the information sheet for the study of health and iodine status of babies (HIBA) and that I have had the opportunity to ask guestions. I understand that taking part is voluntary and that I am free to withdraw at any time without giving a reason, and that my legal rights and medical treatment will not be affected. I understand that I can ask for further information or explanations at any time during the study. **USE OF YOUR INFORMATION** 2. I give permission for authorised individuals from the HIBA team to access information and records collected by the hospital, midwives and health visitors about me and my baby during and after my pregnancy. I give permission for information from the hospital about my pregnancy to be linked to information collected for this study. I understand that relevant sections of information collected in the study will be looked at by authorised individuals from the HIBA team. I give permission for these individuals to have access to these records and to collect, store, analyse and publish information obtained from my taking part in this study. I understand that my personal details will be kept confidential and my name will not be disclosed. 3. I understand that should I withdraw from the study then the information collected so far cannot be erased and may still be used by the researchers. **BLOOD AND URINE SAMPLES** 4. I agree to blood and urine samples being collected around the 12th, 26th and 36th weeks of my pregnancy, and again around 6, 18 and 30 weeks after delivery. **5.** I understand the HIBA team and their research partners in the UK, will use these samples. I understand that the results of individual tests will not be published in any way that reveals my identity. 6. I give permission for the information collected and any spare biological samples to be kept and used for future approved studies regarding health and pregnancy. 7. If I wish to withdraw from the study I agree that these samples may be kept and used, unless I request that they be destroyed. In this case I understand that the research team will make every effort to do so and to ensure that there is no further use of the samples. THYROID ASSESSMENT 8. I agree to a nurse, midwife or doctor assessing the size of my thyroid. I understand that this information may be passed to my GP for further investigation if necessary. Name of participant Date Signature ...... Name of person taking consent Date Signature (if different from researcher) Name of researcher Date Signature